CLINICAL TRIAL: NCT06088537
Title: Isolated Rectal Bleeding in Newborns : Allergic Proctocolitis or Neonatal Colitis Transient - COLON Study
Acronym: COLON
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23-PP-05
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Isolated Rectal Bleedings
Keywords: allergic proctocolitis; neonatal colitis transient; cow's milk protein allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational pilot study evaluating the frequency of cow's milk protein allergic prococolitis in newborns hospitalized in neontal medicine at the university hospital of Nice who presented rectal bleeding.

DETAILED DESCRIPTION:
Inclusion of all newborns in the neonatal medicine department at Nice University Hospital with isolated rectal bleeding.

A note of information and non-opposition will be presented and given to the biological mother. She has the right to object to this study, on her own initiative, at any time.

Collection of data relating to the newborn during hospitalization, the results of the clinical examination and the systematic check-up carried out in accordance with standard practice, and data at discharge.

Follow-up of the newborn to determine the cause of rectal bleeding and therefore the frequency of procolitis allergic to cow's milk proteins.

Prospective observational study of current practices without any intervention.

ELIGIBILITY:
Inclusion Criteria:

1. All newborns ≤ 28 days corrected age or ≤ 44 amenorrhea weeks corrected age hospitalized in neonatal medicine with isolated rectorrhagia;
2. Affiliated to social security ;
3. Presenting isolated rectorrhagia defined as rectorrhagia without hematemesis/ repeated vomiting/ tense or distended abdomen/ apathy/ apnea/ bradycardia or signs of severity (tachycardia, desaturation, poor coloration);
4. After obtaining the biological mother's non-objection;

Exclusion Criteria:

1. All newborns with ulcerative enterocolitis, congenital digestive malformations or rectorrhagia following digestive surgery;
2. Opposition to participation in research involving the human person.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns ≤ 28 days corrected age or ≤ 44 amenorrhea weeks corrected age hospitalized in neonatal medicine with isolated rectorrhagia.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-07-24 (Estimated); Study Completion 2027-07-24 (Estimated)

PRIMARY OUTCOMES:
Number of newborns allergic to cow's milk protein and hospitalized in neonatal medicine at Nice University Hospital with isolated rectorrhagia. | 3 years
  The main objective of this study is to determine the number of newborns presenting real allergic proctocolitis to cow's milk protein among all newborns hospitalised in neonatal medicine who presented with isolated rectal bleeding in order to determine the frequency of this pathology.
  If rectal bleeding disappears when cow's milk proteins are eliminated and reappears when cow's milk proteins are reintroduced, the diagnosis of allergic proctocolitis to cow's milk proteins will be confirmed.
  In other cases, newborns will be considered to have had transient neonatal colitis.
  Then this study will determine the frequency of these two diseases in the population study.

SECONDARY OUTCOMES:
Identify risk factors for developing transient neonatal colitis. | 3 years
  To determine these risk factors, the study will compare the characteristics of newborns with allergic protocolitis to cow's milk proteins with those of newborns with transient neonatal colitis.
  The parameters compared between the two groups will be as follows: gestational age at birth, route of delivery, antibiotic therapy prior to rectal bleeding, type of diet (mother's milk or artificial milk) family history of allergy.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice - Hôpital Archet 2, Nice, Alpes-Mritimes, France

IPD SHARING:
Plan to Share IPD: No